CLINICAL TRIAL: NCT00370097
Title: PD of Hydrofluoroalkane Propellant of Inhaled Fluticasone Propionate Following Administration in Pediatric Subjects 6-12 Months of Age With Asthma
Brief Title: FLOVENT Hydrofluoroalkane (HFA) In 6-12 Month Old Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FAS106533
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Asthma infants FLOVENT spacer
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving HFA (Experimental): Subjects in Session 1 will receive two inhalations of placebo HFA by meter-dose inhaler (MDI) twice daily and in Session 2 subjects will receive two inhalations of fluticasone propionate (FP) HFA MDI 44 mcg twice daily
  Interventions: Drug: FLOVENT (fluticasone propionate) HFA; Drug: Placebo HFA

INTERVENTIONS:
Drug: FLOVENT (fluticasone propionate) HFA — FLOVENT HFA consists of a white to off-white suspension of FP (micronized) in a liquefied hydrofluoroalkane propellant, 1,1,1,2-tetrafluoroethane. Subject will receive FP HFA using an Aerochamber Plus with Infant Mask.
Drug: Placebo HFA — Subjects will receive FP-matched placebo using an Aerochamber Plus with Infant Mask.

SUMMARY:
The purpose of this study is to address an Food Drug and Administration (FDA) request to provide safety data in pre-asthmatic patients, ages 6 months to <12 months, following administration of fluticasone propionate HFA.

DETAILED DESCRIPTION:
A repeat-dose, open-label, 2-session study to assess the systemic exposure to, and pharmacodynamics of, fluticasone propionate HFA inhalation aerosol 88mcg administered twice-daily for 28 days delivered via an MDI and valved holding chamber with infant facemask to subjects ages 6 months to <12 months who have experienced 2 or more wheezing episodes in the preceding 6 months

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have experienced 2 or more wheezing episodes in the previous 6 months.
* Subjects may not have taken any corticosteroids in the 4 weeks prior to dosing
* Parents/guardians should be able to read and comprehend diary information collected throughout the study
* Parents must be able to demonstrate the ability to use the facemask and spacer used to administer study drug

Exclusion criteria:

* Subjects who weigh less than 7 kg
* Subjects who are taking any drugs that inhibit or induce the cytochrome P450 isoform
* Any parents who have a history of psychiatric disease, intellectual deficiency, substance abuse that would compromise the validity of the consent

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2006-08-30 (Actual); Primary Completion 2007-04-12 (Actual); Study Completion 2007-04-12 (Actual)

PRIMARY OUTCOMES:
Serum cortisol weighted mean(0-12h) | throughout the study

SECONDARY OUTCOMES:
Serum cortisol Cmin FP Cmaxss, AUClast and tmaxss Adverse events | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study FAS106533 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/FAS106533?search=study&search_terms=FAS106533#rs
- Available data/document: Clinical Study Report: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FAS106533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register